CLINICAL TRIAL: NCT04053049
Title: Advancing Nutritional Science for Children With Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: NASPGHAN Foundation (Other Government)
Responsible Party: Principal Investigator, Bruno Chumpitazi, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H-44307
Record Dates: First submitted 2019-05-03; First posted 2019-08-12 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Each subject will receive 4 meals of different composition.
Who Masked: Participant, Investigator
Masking Description: Meals will be provided in a randomized fashion with only the metabolic research unit kitchen (which prepares the meals) knowing what is being provided to the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High fat/ Semi-solid (Active Comparator): Subject will receive a high fat/semi-solid meal.
  Interventions: Other: Diet
- High carbohydrate/ Semi-solid (Active Comparator): Subject will receive a high carbohydrate/semi-solid meal.
  Interventions: Other: Diet
- High fat/ solid (Active Comparator): Subject will receive a high fat/solid meal.
  Interventions: Other: Diet
- High carbohydrate/ solid (Active Comparator): Subject will receive a high carbohydrate/solid meal.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Meals composed of either high fat vs. high carbohydrate and semi-solid vs. solid

SUMMARY:
This study evaluates four different meals and how they induce gastrointestinal symptoms in children with functional dyspepsia. All subjects will receive each meal and rate their gastrointestinal symptoms during each meal.

DETAILED DESCRIPTION:
Food can often exacerbate gastrointestinal symptoms in adults and children with functional dyspepsia. However, it is unclear which foods exacerbate symptoms more than others.

Children with post-prandial distress functional dyspepsia will receive four different meals with variables being: semi-solid vs. solid and high fat vs high carbohydrate. At the time of ingestion and for up to 3 hours after each meal, subjects will rate their gastrointestinal symptoms. Comparisons of symptom onset and severity will be made for each meal.

Enrolled subjects will have undergone previous gastrointestinal evaluations: gastric emptying study and/or upper endoscopy. In addition, subjects will complete psychosocial measures: Behavioral Assessment for Children-3, childhood somatization inventory.

The first goal is to compare the severity of gastrointestinal symptoms with different composition and consistency meals. The second goal is to correlate the severity of postprandial gastrointestinal symptoms to psychosocial distress, gastric neuromotor function (emptying and accommodation), and duodenal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Rome IV Functional Dyspepsia with post-prandial distress
* Previously completed normal upper endoscopy with duodenal biopsies and/or previously completed a gastric emptying scintigraphy study

Exclusion Criteria:

* Previous abdominal surgery
* Current or previous formal psychiatric diagnosis (e.g. anxiety disorder) requiring therapy or psychotropics
* Serious chronic medical condition requiring regular medical care
* Allergy to meal components to be ingested during the study
* On specialized diet required for a medical condition
* Pregnancy
* Inability to eat by mouth

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Dyspepsia Symptom Severity | up to 16 weeks
  Change from baseline gastrointestinal symptoms using total visual analogue scale score

SECONDARY OUTCOMES:
Dyspepsia Symptom Onset | up to 16 weeks
  Time to maximum symptom severity
Duodenal inflammation | up to 16 weeks
  Previously obtained duodenal mucosal biopsies will be re-evaluated for eosinophils and mast cells
Gastric retention | up to 16 weeks
  Gastric retention values will be captured from a previously completed 4-hour gastric emptying scintigraphy study
Psychosocial distress | up to 16 weeks
  Anxiety, Depression, and Somatization will be determined using Behavioral Assessment for Children-3 (t-scores for anxiety and depression) and Children's Somatization Inventory Score (total score).
Gastric accommodation | up to 16 weeks
  Gastric accommodation will be determined from a previously completed 4-hour gastric scintigraphy study using analysis of the time zero image.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Chumpitazi, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No